CLINICAL TRIAL: NCT06353529
Title: Effect of Sphenopalatine Ganglion Block with Bupivacaine on Postoperative Pain in Patients Undergoing Endoscopic Pituitary Adenoma Resection
Brief Title: Postop Pain Management in Pituitary Tumour Patients
Acronym: POPPY
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17065
Record Dates: First submitted 2024-03-26; First posted 2024-04-09 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-04

CONDITIONS: Pituitary; Pain, Postoperative
Keywords: Nerve block; Bupivacaine; Sphenopalatine Ganglion
MeSH Terms: conditions — Pituitary Diseases; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Bupivacaine injection (Experimental): This group will receive bilateral injection of 0.5% bupivacaine with 1:200,000 epinephrine using a 20G needle and comprising 2mL of fluid on each side (4mL total) into the sphenopalatine ganglion.
  Interventions: Drug: Bupivacaine-Epinephrine 0.5%-1:200,000 Injectable Solution
- Placebo Control (Placebo Comparator): This group will receive bilateral injection of 0.9% saline solution using a 20G needle and comprising 2mL of fluid on each side (4mL total) into the sphenopalatine ganglion.
  Interventions: Drug: Placebo
- Sham - no injection (Sham Comparator): Participants randomized to this arm will not receive any additional study injections and will undergo the current standard procedure for patients undergoing endoscopic endonasal surgery.
  Interventions: Drug: Sham Comparator

INTERVENTIONS:
Drug: Bupivacaine-Epinephrine 0.5%-1:200,000 Injectable Solution — 2mL injection bilateral (4mL total) of 0.5% bupivacaine with 1:200,000 epinephrine solution, 20G needle, sterile, sphenopalatine ganglion; nerve block
  Arms: Bupivacaine injection
Drug: Placebo — 2mL injection bilateral (4mL total) 0.9% saline solution, 20G needle, sterile, sphenopalatine ganglion; nerve block
  Arms: Placebo Control
Drug: Sham Comparator — Participants receive no additional study injections
  Arms: Sham - no injection

SUMMARY:
To assess the benefit of using an additional nerve block during minimally invasive pituitary surgery, to improve pain management after surgery. The medication (Bupivacaine) or a placebo (saline) will be injected during surgery and patients will be asked about their level of pain at multiple time points in the first 24 hours following surgery. Some patients will be randomized to a third, sham group that do not receive any additional injection. The aim is to improve patient outcomes and reduce the need for pain medication after surgery.

DETAILED DESCRIPTION:
To further improve the quality of the early postoperative course, the investigators propose the use of the sphenopalatine ganglion (SPG) block (SPGB) for pain management in the context of an enhanced recovery after surgery (ERAS) protocol for minimally invasive (MIS) endoscopic transsphenoidal pituitary surgery. The SPG is the main sensory innervation to the nasal mucosa, and several studies have shown the analgesic efficacy of SPGB following sinus surgery and showed positive results for endoscopic sinus surgery. However, there is limited research on the use of SPGB in the context of pituitary surgery.

In this randomized placebo-controlled trial, the investigators aim to assess the benefit of SPGB with bupivacaine in addition to multimodal general anesthesia on pain management, after MIS pituitary surgery. The results of the trial will provide valuable insights into the potential benefits of SPGB and its optimal use for pituitary surgery.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (18 yrs or older)
* undergoing endonasal pituitary adenoma resection

Exclusion Criteria:

* Patients with pre-existing chronic pain conditions requiring antidepressants (serotonin reuptake inhibitors), benzodiazepines, gabapentin, or opioid drugs
* contraindications to the performance of SPGB such as known allergy to used medications
* chronic alcohol abuse
* uncontrolled systemic arterial hypertension
* severe kidney or liver diseases
* cardiomyopathies or sustained cardiac arrhythmias (permanent paroxystic atrial fibrillation or other sustained supraventricular rhythmic anomalies)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain score | through study completion, approximately 1 year
  Pain score, measured by visual analog scale (scale of 0-10) at 6, 12 and 24 hours post-op

SECONDARY OUTCOMES:
Post-operative bleeding | through study completion, approximately 1 year
  amount of post-op bleeding (mL) in first 24 hours
Post-operative complications | through study completion, approximately 1 year
  record presence of post-op nausea/vomiting, headache, sore throat, difficulty swallowing in first 24 hours
Analgesic requirement | through study completion, approximately 1 year
  List and dose of analgesics administered to patient in first 24 hours or time of discharge, whichever comes first
Length of stay | through study completion, approximately 1 year
  Length of hospital stay in hours

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Kesava Reddy, MD, Principal Investigator — Hamilton Health Sciences Corporatin
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Patient data will be de-identified and the data will be analyzed as a whole before becoming available to other researchers.
  De-identified IPD may be shared with other researchers if necessary based on occurrence of adverse events occurrence, circumstantial findings, etc.

REFERENCES:
- [Background] Morisse M, Rysman B, Szymanski C, Fackeure R, Mouawad F, Mortuaire G. A randomized placebo-controlled trial assessing sphenopalatine ganglion block in endoscopic sinus surgery. Int Forum Allergy Rhinol. 2021 Sep;11(9):1384-1386. doi: 10.1002/alr.22804. Epub 2021 May 19. No abstract available. PMID 34013619
- [Background] Rezaeian A, Hashemi SM, Dokhanchi ZS. Effect of Sphenopalatine Ganglion Block With Bupivacaine on Postoperative Pain in Patients Undergoing Endoscopic Sinus Surgery. Allergy Rhinol (Providence). 2019 Jan 23;10:2152656718821282. doi: 10.1177/2152656718821282. eCollection 2019 Jan-Dec. PMID 30719401
- [Background] Kim DH, Kang H, Hwang SH. The Effect of Sphenopalatine Block on the Postoperative Pain of Endoscopic Sinus Surgery: A Meta-analysis. Otolaryngol Head Neck Surg. 2019 Feb;160(2):223-231. doi: 10.1177/0194599818805673. Epub 2018 Oct 9. PMID 30296912
- [Background] Kesimci E, Ozturk L, Bercin S, Kiris M, Eldem A, Kanbak O. Role of sphenopalatine ganglion block for postoperative analgesia after functional endoscopic sinus surgery. Eur Arch Otorhinolaryngol. 2012 Jan;269(1):165-9. doi: 10.1007/s00405-011-1702-z. Epub 2011 Jul 8. PMID 21739090
- [Background] Wang P. The efficacy of sphenopalatine ganglion block for pain management after endoscopic sinus surgery: a meta-analysis of randomized controlled studies. Eur Arch Otorhinolaryngol. 2021 Aug;278(8):2681-2687. doi: 10.1007/s00405-020-06484-9. Epub 2021 Jan 3. PMID 33388988